CLINICAL TRIAL: NCT03339141
Title: Comparison of Intubating Conditions in 25° Head-up Position and Strict Supine
Acronym: InSizeS25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-361; 2016-A02078-43 (Other: 2016-A02078-43)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Intubation; Intratracheal
Keywords: Intubation conditions; Anaesthetic techniques; Laryngoscopy

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine position (Placebo Comparator): Patients are placed in the supine position at 0° from arrival in the room until intubation
  Interventions: Procedure: Intubation position
- 25° head-up position (Active Comparator): Patients are placed in the 25° head-up position (half-seat or whole body proclive) from arrival in the room until intubation.
  Interventions: Procedure: Intubation position

INTERVENTIONS:
Procedure: Intubation position — The investigators assess two different patient's intubation position : supine position and 25° head-up position looking at the intubation score (POGO score).

SUMMARY:
Tracheal intubation, particularly before surgery, is traditionally done in supine position. It was shown in the general population and in obese patients in particular, that the pre-oxygenation in a 25° head-up position provided a better efficiency of the pre-oxygenation and an apnea time longer. This position would also allow for better intubation conditions in direct laryngoscopy.

The investigators intend to assess two different patient's intubation position : supine position and 25° head-up position

DETAILED DESCRIPTION:
Randomization assigned in random block, stratification by operator (20 patients per operator, 10 in each group).

Interim analysis every 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* - patients scheduled for various surgeries requiring general anesthesia with curare, with intubation of the trachea, eligible for intubation by direct laryngoscopy.
* > 18 years
* patients with social security

Exclusion Criteria:

* Emergency surgery.
* Patient who requiring rapid sequence induction.
* Intubation without curare.
* Expected difficult intubation with planned modification of the intubation protocol (i. e. intubation under fibroscopy, airtrach or videolaryngoscopy)
* Patient with a history of epilepsy, pulmonary or cardiovascular disease (including ischemic heart disease, symptomatic asthma or obstructive pulmonary disease).
* Patient with mask phobia.
* BMI> 30kg / m2
* Patient who are refusing to take part.
* Patient protected major, minor, pregnant women, patients deemed incapable of giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
POGO score | at day 1
  valid score observed by the anesthetist performing intubation at the time of intubation. POGO score means Percentage of Glottic Opening : from 0% (none visualization of the glottic opening, worst result) to 100% (complete visualization of the glottic opening, best result), from the anterior curvature of the vocal cords to the interarytenoid node, between the posterior cartilage

SECONDARY OUTCOMES:
Cormack-Lehane grade | at day 1
  another valid score observed by the anesthetist performing intubation at the time of intubation. It classifies views obtained by direct laryngoscopy based on the structures seen. From 1 (best result) to 4 (worst result). 1 : full view of glottis (POGO 100%) / 2 : partial view of glottis / 3 : only epiglottis seen, none of glottis seen (POGO 0%) / 4 : Neither glottis nor epiglottis seen (POGO 0%).
Intubation operator's comfort | at day 1
  visual analog scale about the operator's comfort during intubation. It's a subjective score. It's an evaluation of the comfort of the intubation position from 0 to 10, where 0 is a total discomfort, a painful, very uncomfortable position and 10 is an optimal, very comfortable position.
Episodes of desaturation and episodes of hypotension | at ady 1
  SpO2 <90% or MAP <65mmHg or drop> 20% of the patient's baseline SBP
Mechanical complications of intubation: | at day 1
  laryngeal pain, hoarseness, upper airway trauma
Patient height | at day 1
  at the tragus of the ear during intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne BAZIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (6):
- France (6):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Pôle Santé République, Clermont-Ferrand
  - Centre Hospitalier Alpes-Léman, Contamine-sur-Arve
  - Polyclinique Saint Odilon, Moulins
  - Hôpital Saint-Louis / AP-HP, Paris
  - Hôpital Nord-Ouest, Villefranche-sur-Saône

REFERENCES:
- [Derived] Falempin AS, Pereira B, Binakdane F, Bazin JE, Smirdec M. Investigator-initiated, multicentre, open-label, two-arm, randomised controlled trial comparing intubating conditions in 25 degrees head-up position and supine: the InSize25 study protocol. BMJ Open. 2019 Nov 3;9(11):e029761. doi: 10.1136/bmjopen-2019-029761. PMID 31685496